CLINICAL TRIAL: NCT00603434
Title: Double-Blind, Placebo-Controlled Assessment of Potential Interactions Between Intravenous Methamphetamine and Osmotic-Release Methylphenidate (OROS-MPH)
Brief Title: Safety Assessment of Potential Interactions Between IV Methamphetamine and Osmotic-Release Methylphenidate (OROS-MPH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Liza Gorgon, NIDA
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NIDA-CPU-Methylphenidate-0001
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-03

CONDITIONS: Methamphetamine Dependence; Methamphetamine Abuse
Keywords: Methamphetamine
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Osmotic-Release Methylphenidate
  Interventions: Drug: OROS-MPH
- 2 (Experimental): Osmotic-Release Methylphenidate
  Interventions: Drug: OROS-MPH
- 3 (Experimental): Osmotic-Release Methylphenidate
  Interventions: Drug: OROS-MPH

INTERVENTIONS:
Drug: OROS-MPH — 18 mg bid on days 1 and 2
  Other Names: Concerta
  Arms: 1
Drug: OROS-MPH — 27mg bid on days 3 and 4
  Other Names: Concerta
  Arms: 2
Drug: OROS-MPH — 35 mg bid on days 5-9
  Other Names: Concerta
  Arms: 3

SUMMARY:
This is a human inpatient clinical pharmacology study to assess potential interactions between intravenous (i.v.) methamphetamine infusion and oral osmotic release methylphenidate (OROS-MPH). The primary objective of this study is to determine the safety of the OROS-MPH concurrent with i.v. d-methamphetamine infusions of 15 mg and 30 mg. Safety outcome measures include cardiovascular responses [heart rate (HR), blood pressure (BP), and electrocardiograph (ECG) measurements], oral temperature, adverse events (AEs), and clinical laboratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Be volunteers who meet DSM-IV criteria for methamphetamine abuse or dependence determined using a Mini-International Neuropsychiatric Interview (MINI) and be non-treatment seeking at time of study and have a positive urine test for methamphetamine (greater than or = to 500 ng/mL) during screening.
* Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
* Have a negative urine test for methamphetamine and other drugs of abuse (opiates, cocaine, and benzodiazepines) after clinic intake before the first infusion session.
* Have a history and physical examination that demonstrate no clinically significant contraindication for participating in the study, in the judgment of the admitting physician and the site Principal Investigator
* Have vital signs as follows: resting heart rate between 45 and 100 bpm, systolic BP below 140 mm Hg and diastolic BP below 90 mm Hg.
* Have electrolytes (Na, K, Cl, HCO3) and hematocrit that is clinically normal (+/- 10% of laboratory limits).
* Have liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) less than three times the upper limit of normal.
* Have kidney function tests (creatinine and BUN) less than twice the upper limit of normal.
* Have an ECG performed that demonstrates sinus rhythm between 45 and 100 beats per minute (bpm), normal conduction, and no clinically significant arrhythmias.
* Be able to swallow whole tablets of OROS-MPH due to the controlled release formulation.
* If female, have a negative pregnancy test and agree to use one of the following methods of birth control, or be postmenopausal, have had a hysterectomy or have been sterilized. Birth control must be in effect starting at least 7 days (14 days for hormone-based methods used alone) prior to clinic intake, and should extend at least until the last follow-up visit.

Exclusion Criteria:

* Please contact site for more information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety of the OROS-MPH concurrent with d-methamphetamine infusions. | Daily

SECONDARY OUTCOMES:
Plasma concentrations | Screen, day 2, day 10

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, MD, PhD, Principal Investigator — University of Cincinnati; Edward Sellers, MD, PhD, Principal Investigator — Ventana Clinical Research Corporation
Locations (2):
- Cincinnati Addiction Research Center, Cincinnati, Ohio, United States
- Ventana Clinical Research Corporation, Toronto, Ontario, Canada